CLINICAL TRIAL: NCT03506360
Title: Phase 2 Trial of Pembrolizumab, Ixazomib, and Dexamethasone for Relapsed Multiple Myeloma
Brief Title: Pembrolizumab, Ixazomib Citrate, and Dexamethasone in Treating Patients With Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1782; NCI-2018-00590 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1782 (Other: Mayo Clinic in Rochester); 17-008639 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2018-04-11; First posted 2018-04-24 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Recurrent Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; ixazomib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ixazomib citrate, pembrolizumab, dexamethasone) (Experimental): Patients receive ixazomib citrate PO on days 1, 8, 15, 29, 36, 43, 57, 64, and 71 and pembrolizumab IV over 30 minutes on days 1, 22, 43, 64. Patients also receive dexamethasone PO on days 1, 8, 15, 29, 36, 43, 57, 64, and 71. Cycles with dexamethasone repeat every 84 days for up to 1 year and cycles with ixazomib citrate and pembrolizumab repeat every 84 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Drug: Ixazomib Citrate; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; Ninlaro
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab works when given together with ixazomib citrate and dexamethasone in treating patients with multiple myeloma that has come back (relapsed). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Ixazomib citrate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pembrolizumab together with ixazomib citrate and dexamethasone may work better in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the overall response rate (>= partial response [PR]) of pembrolizumab in combination with standard doses of ixazomib citrate (ixazomib) and dexamethasone, in patients with relapsed symptomatic multiple myeloma (MM).

SECONDARY OBJECTIVES:

I. To determine the >= very good partial response (VGPR) and complete response (CR) rate of pembrolizumab added to standard doses of ixazomib and dexamethasone in relapsed myeloma.

II. To determine the progression free survival and overall survival among patients with relapsed MM following treatment with the combination of pembrolizumab, ixazomib and dexamethasone.

III. To determine the toxicities associated with pembrolizumab added to standard doses of ixazomib and dexamethasone in patients with relapsed MM.

CORRELATIVE RESEARCH:

I. PDL-1 expression on myeloma cells and non-tumor cell compartments from the bone marrow will be assessed at baseline.

II. Measures of T-cell activation/exhaustion will be assessed at baseline and after cycle 1 and cycle 3.

III. Natural killer (NK) cell function and numbers will be evaluated at baseline and after cycle 1 and cycle 3.

OUTLINE:

Patients receive ixazomib citrate orally (PO) on days 1, 8, 15, 29, 36, 43, 57, 64, and 71 and pembrolizumab intravenously (IV) over 30 minutes on days 1, 22, 43, 64. Patients also receive dexamethasone PO on days 1, 8, 15, 29, 36, 43, 57, 64, and 71. Cycles with dexamethasone repeat every 84 days for up to 1 year and cycles with ixazomib citrate and pembrolizumab repeat every 84 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months until progressive disease, and then every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed, symptomatic multiple myeloma by International Myeloma Working Group (IMWG) diagnostic criteria for multiple myeloma
* Age >= 18 years
* Calculated creatinine clearance (using Cockcroft-Gault equation below) >= 30 mL/min (obtained =< 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1000/mm^3 (obtained =< 14 days prior to registration)
* Platelet count >= 75000/mm^3; Note: Platelet transfusion is not allowed =< 3 days prior to registration (obtained =< 14 days prior to registration)
* Hemoglobin >= 8.0 g/dL (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 14 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN (obtained =< 14 days prior to registration)
* Must have relapsed or refractory disease after treatments including three therapies: proteasome inhibitors, immunomodulatory imide drugs (IMiDs), and anti-CD38 antibody
* Measurable disease of multiple myeloma as defined by at least ONE of the following:

  * Serum monoclonal protein >= 1.0 g/dL
  * >= 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, or 1
* Provide informed written consent
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Willing to follow strict birth control measures;

  * Female patients: If they are of childbearing potential, agree to one of the following:

    * Practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 120 days after the last dose of study drug, AND must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
  * Male patients: even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

    * Agree to practice effective barrier contraception during the entire study treatment period and through 120 days after the last dose of study drug, OR
    * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* Willing to provide bone marrow and blood samples for planned research

Exclusion Criteria:

* Myeloma disease that is refractory to ixazomib treatment
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include early stage cancers (carcinoma in situ or stage 1) treated with curative intent, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer, or in situ breast cancer that has undergone potentially curative therapy
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Other co-morbidity which would interfere with patient's ability to participate in trial, e.g. uncontrolled infection, uncompensated heart or lung disease
* Other concurrent chemotherapy, or any ancillary therapy considered investigational =< 14 days prior to study registration; NOTE: Bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* Peripheral neuropathy >= grade 3 on clinical examination or grade 2 with pain during the screening period
* Major surgery =< 14 days prior to study registration
* Radiotherapy =< 14 days prior to registration; NOTE: If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of study drugs
* Participation in any other clinical trials with other investigational agents not included in this trial =< 21 days prior to registration
* Has active autoimmune disease that has required systemic treatment =< 2 years prior to study registration (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs);

  * NOTE: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has a known history of interstitial lung disease
* Has an active infection requiring systemic therapy
* Has a history of current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has a known history of active TB (Bacillus tuberculosis)
* Has received a live vaccine =< 30 days prior to study registration
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Allogeneic hematopoietic stem cell transplant
* Systemic treatment with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort =< 14 days prior to registration
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2020-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lin, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ixazomib Citrate, Pembrolizumab, Dexamethasone)
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This study is permanently closed early due to slow accrual.
Groups:
- Treatment (Ixazomib Citrate, Pembrolizumab, and Dexamethasone): Patients receive ixazomib citrate PO on days 1, 8, 15, 29, 36, 43, 57, 64, and 71 and pembrolizumab IV over 30 minutes on days 1, 22, 43, 64. Patients also receive dexamethasone PO on days 1, 8, 15, 29, 36, 43, 57, 64, and 71. Cycles with dexamethasone repeat every 84 days for up to 1 year and cycles with ixazomib citrate and pembrolizumab repeat every 84 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
Arm/Group | Treatment (Ixazomib Citrate, Pembrolizumab, and Dexamethasone)
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 67 [41 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Percentage
Description: Defined as a partial response or better noted as the objective status on two consecutive evaluations. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.
Time Frame: Up to 9 months
Measure: Number (90% Confidence Interval); unit: percentage of responders
Arm/Group | Treatment (Ixazomib Citrate, Pembrolizumab, and Dexamethasone)
Number analyzed (Participants) | 13
percentage of responders | 0.077 [0.004 to 0.322]

2. Secondary Outcome: >= Very Good Partial Response (VGPR) Response Percentage With Pembrolizumab Added to Ixazomib Citrate and Dexamethasone
Description: Will be estimated by the number of patients who achieve a VGPR, complete response (CR), or stringent complete response (sCR) at any time divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success rate will be calculated.
Time Frame: Up to 9 months
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Treatment (Ixazomib Citrate, Pembrolizumab, and Dexamethasone)
Number analyzed (Participants) | 13
percentage of responders | 0 [NA to NA] — No events occurred, intervals are incalculable

3. Secondary Outcome: Complete Response Percentage With Pembrolizumab Added to Ixazomib Citrate and Dexamethasone
Description: Will be estimated by the number of patients who achieve a CR or sCR at any time divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success rate will be calculated.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Treatment (Ixazomib Citrate, Pembrolizumab, and Dexamethasone)
Number analyzed (Participants) | 13
percentage of responders | 0 [NA to NA] — No events occurred, intervals incalculable

4. Secondary Outcome: Survival Time
Description: The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Ixazomib Citrate, Pembrolizumab, and Dexamethasone)
Number analyzed (Participants) | 13
Months | 9 [3 to NA] — No enough events occurred to obtain an upper limit.

5. Secondary Outcome: Progression-free Survival
Description: The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Ixazomib Citrate, Pembrolizumab, and Dexamethasone)
Number analyzed (Participants) | 13
Months | 1.6 [0.7 to 2.8]

6. Secondary Outcome: Incidence of Adverse Events
Description: Graded according National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.
Time Frame: Up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ixazomib Citrate, Pembrolizumab, and Dexamethasone)
Number analyzed (Participants) | 13
Participants | 13

7. Other Pre Specified Outcome: PDL-1 Expression on Myeloma Cells and Non-tumor Cell Compartments From the Bone Marrow
Description: Each measure will be summarized descriptively by median, minimum (min), maximum (max) and interquartile range.
Time Frame: Baseline
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Markers of T-cell Activation and Exhaustion
Description: Will be summarized descriptively by median, min, max, and interquartile range at each time point. Patterns over time will be summarized by absolute difference or relative change. Changes across time will be assessed using paired analyses, including Wilcoxon signed rank tests. Jitplots will be used to visually examine differences between groups for continuous factors.
Time Frame: Baseline up to Cycle 3 (84 days - each Cycle is 28 days)
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Natural Killer Cell Function and Numbers
Description: as for outcome 8
Time Frame: Baseline up to Cycle 3 (84 days - each Cycle is 28 days)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Treatment (Ixazomib Citrate, Pembrolizumab, and Dexamethasone)
All-Cause Mortality (participants affected / at risk) | 6/13
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ixazomib Citrate, Pembrolizumab, and Dexamethasone) (N=13)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ixazomib Citrate, Pembrolizumab, and Dexamethasone) (N=13)
Anemia (Blood and lymphatic system disorders) | 6 (9)
Constipation (Gastrointestinal disorders) | 6 (19)
Diarrhea (Gastrointestinal disorders) | 3 (10)
Nausea (Gastrointestinal disorders) | 5 (10)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 12 (40)
Creatinine increased (Investigations) | 7 (22)
Lymphocyte count decreased (Investigations) | 6 (19)
Lymphocyte count increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 3 (4)
Platelet count decreased (Investigations) | 11 (32)
White blood cell decreased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT03506360/Prot_SAP_000.pdf